CLINICAL TRIAL: NCT01503203
Title: Physical Virtual Training Effectiveness on Nonspecific Chronic Low Back Pain, Body Balance, Functional Autonomy and Mood of Older Women
Brief Title: Physical Virtual Training for Older Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Gama Filho (Other)
Responsible Party: Principal Investigator, Renato Sobral Monteiro Junior, Clinical Professor, Universidade Gama Filho
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RSMJ20112
Record Dates: First submitted 2011-12-16; First posted 2012-01-02 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Low Back Pain
Keywords: Older; virtual systems; low back pain; postural balance
MeSH Terms: conditions — Low Back Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wii Group (Experimental): This group will do the same training of the Prime Group. However will do also Physical Virtual Training using Nintendo Wii and Wii Balance Board. The physical virtual training going to applied during thirty minutes.
  Interventions: Other: Physical Virtual Training; Other: Strength Training; Other: Core Training
- Prime Group (Active Comparator): This group will do strength exercises and core training.
  Interventions: Other: Strength Training; Other: Core training

INTERVENTIONS:
Other: Strength Training — It will be does three times per week. The exercises are: squat, single leg squat, leg extension, leg curl, chair adductor, chair abductor and double plantar flexion.
  Other Names: Resistance training
  Arms: Prime Group
Other: Core training — Exercises for trunk stabilization. Will be lateral, front and back bridges. It will be does three times per week with three sets between fifteen and third seconds.
  Arms: Prime Group
Other: Physical Virtual Training — The video game (Nintendo Wii and Wii Balance Board) will used for intervention. After strength and core training will be applied the physical virtual training during thirty minutes. Tho total time session for the Wii Group will be 110 minutes.
  Arms: Wii Group
Other: Strength Training — It will be does three times per week. The exercises are: squat, single leg squat, leg extension, leg curl, chair adductor, chair abductor and double plantar flexion.
  Other Names: Resistance training
  Arms: Wii Group
Other: Core Training — Exercises for trunk stabilization. Will be lateral, front and back bridges. It will be does three times per week with three sets between fifteen and third seconds.
  Arms: Wii Group

SUMMARY:
The purpose of this study will be assess the effectiveness of the physical virtual training on nonspecific chronic low back pain, body balance, functional autonomy and mood of older women. Two groups will be formed. One will do strength exercises and core training. The other group will do the same exercises more virtual activities with Nintendo Wii. Will be measure pre and post-intervention of the responses already shown above.

ELIGIBILITY:
Inclusion Criteria:

* subjects with nonspecific chronic low back pain
* patients without involvement in regular exercise program

Exclusion Criteria:

* patients not recommended for physical exercise (Physical Activity Readiness Questionnaire PAR-Q)
* trunk surgery
* cancer
* injuries in lower extremity
* neurological or vestibular disease

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-04 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Pain | up to 8 weeks
  The low back pain will be assessed with numeric pain scale two times (pre and post-intervention).

SECONDARY OUTCOMES:
Body Balance | up to 8 weeks
  The body balance will be assessed with Wii Balance Board two times (pre and post-intervention).
Functional autonomy | up to 8 weeks
  The functional autonomy will be assessed with sit-to-stand test pre and post-intervention.
Mood | up to 8 weeks
  The mood will be assessed with Profile of Mood State (POMS) two times (pre and post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Elirez B da Silva, Doctor, Study Director — Gama Filho University
Locations (1):
- Fisioprime Clinical of Physiotherapy, Rio de Janeiro, Rio de Janeiro, Brazil